CLINICAL TRIAL: NCT06022510
Title: Safety and Efficacy of Fetoscopes Used in Fetoscopic Selective Laser Photocoagulation for Complicated Monochorionic-Diamniotic Pregnancies
Brief Title: Safety and Efficacy of Fetoscopes Used in Fetoscopic Selective Laser Photocoagulation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: These fetoscopes have obtained FDA approval under Karl Storz's existing HDE (H040005) for their fetoscopy instrument set. No participants were enrolled as we did not receive the fetoscopes until early 2025 and the IDE is closed as of April 2025.
Sponsor: Michael A Belfort (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Michael A Belfort, Chairman and Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-53644
Record Dates: First submitted 2023-08-22; First posted 2023-09-05 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Twin Monochorionic Diamniotic Placenta
Keywords: twin-twin transfusion syndrome; TTTS; twin anemia polycythemia sequence; TAPS; selective intrauterine growth restriction; sIUGR
MeSH Terms: conditions — Fetofetal Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Fetoscopes for Selective Laser Photocoagulation (Experimental): Single arm study. All patients will undergo selective laser photocoagulation with the use of the fetoscopes in this study.
  Interventions: Device: Fetoscopy Sets for Anterior and Posterior Placentas

INTERVENTIONS:
Device: Fetoscopy Sets for Anterior and Posterior Placentas — Patients who choose to undergo fetoscopic surgery for a complicated monochorionic-diamniotic pregnancy will be offered participation in this study. All patients will undergo selective laser photocoagulation with the use of the fetoscopes in this study.
  Other Names: Karl Storz Miniature Straight Forward Telescope 0 Degrees Set - Straight or 11506 AAK; Karl Storz Miniature Straight Forward Telescope 0 Degrees Set - Curved or 11508 AAK

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the investigational fetoscopes used in patients undergoing fetoscopic selective laser photocoagulation for complicated monochorionic-diamniotic pregnancies.

DETAILED DESCRIPTION:
All patients who choose to undergo fetoscopic selective laser photocoagulation (S-PLC) at Texas Children's Fetal Center will be offered participation in this research study by study investigators. Description of study rationale and design and a focused interview by the study coordinator to afford potential participants a formal opportunity to examine what they have learned about the research study in the course of their evaluation and discuss how they feel about enrolling in the research study. Once the patient is deemed eligible the informed consent process will be reviewed. If patients elect to participate in the study, informed consent will be obtained, and patients provided a copy of the signed consent.

Fetoscopic Procedure: Selective laser photocoagulation (S-PLC) is standard of care for the treatment of complicated monochorionic twin pregnancies and will be performed with the same technique in this study as it is with the use of the currently approved fetoscopes. In the majority of cases, in utero access has been achieved using a small percutaneous incision under ultrasound guidance with the instruments inserted through the maternal abdomen, uterine wall and into the recipient fetus' gestational sac. The fetoscope is then used to "map" the placental vascular pattern. Communicating vessels between the fetuses are ablated using laser energy via a 400-600 micron laser fiber that has been introduced through the instrument channel of the operating sheath. Intravenous sedation with local anesthesia at the site of insertion has been found to provide sufficient maternal anesthesia for the procedure. At the completion of the S-PLC, the excess amniotic fluid in the recipient twin's sac is removed to achieve a normal volume.

Follow-Up: The investigators will follow patients for the immediate post-procedure period (until they leave the OR).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible and elect to undergo fetoscopic selective laser photocoagulation for the treatment of complicated monochorionic-diamniotic pregnancies.

Exclusion Criteria:

* Patients who do not elect to undergo fetoscopic laser photocoagulation for treatment of complicated monochorionic-diamniotic pregnancies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Immediate Post-Procedure Period (from surgery start until surgery finish)
  Number of adverse events associated with the investigational device.
Number of device defects, malfunctions, or failures | Immediate Post-Procedure Period (from surgery start until surgery finish)
  Number of device defects, malfunctions, or failures and whether the device performed as intended.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Belfort, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital - Pavilion for Women, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No